CLINICAL TRIAL: NCT07042893
Title: Echocardiographic Assessment of Right Ventricular Function After Pulmonary Resection
Brief Title: Effects of Pulmonary Resection on Right Ventricular Function
Status: Recruiting | Type: Observational
Sponsor: Çağrı Özdemir (Other)
Responsible Party: Sponsor-Investigator, Çağrı Özdemir, asst. prof., Gazi University
Organization: Gazi University (Other)
Other Study IDs: 2024 - 1160
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Resection; Right Ventricular Function; Echocardiography; Cardiothoracic Anesthesia
Keywords: pulmonary resection; right ventricular function; echocardiography; cardiothoracic anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: In this study, a single group (Group 1) will be defined, and patients scheduled for lung resection who agree to participate will be included.

SUMMARY:
Lung resection is associated with high postoperative morbidity and mortality and leads to a significant long-term decrease in functional capacity, particularly due to cardiorespiratory complications. One of the contributing factors to this functional decline is the postoperative reduction in right ventricular function. Due to the anatomical proximity and interactions, right ventricular function is evaluated by echocardiography following lung resection. The pulmonary artery pressure (PAP)/tricuspid annular plane systolic excursion (TAPSE) ratio is a parameter that provides a more comprehensive assessment of right heart function by evaluating both right ventricular systolic function and pulmonary artery pressure. In this study, investigators aimed to evaluate changes in right heart function by performing preoperative and postoperative echocardiographic assessments in participants undergoing lung resection, focusing on PAP/TAPSE ratios.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 80 years

ASA classification I-III

Patients scheduled to undergo lung resection in thoracic surgery

Exclusion Criteria:

Patients with arrhythmia

Patients using antiarrhythmic drugs

Patients with renal failure requiring hemodialysis

Patients with a history of previous lung surgery

Patients with valvular heart disease

Patients with a history of angina pectoris or myocardial infarction within the past month

Patients with FEV1/FVC ratio below 60%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 80 years scheduled to undergo lung resection surgery.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic Assessment: TAPSE/PAP Ratio | 24 hours preoperatively and on postoperative day 2
  Patients will be evaluated by echocardiography 24 hours before surgery and on the second postoperative day, and the TAPSE/PAP ratio will be recorded in mm/mmHg.
Echocardiographic Assessment: Tricuspid Annular Plane Systolic Excursion (TAPSE) | 24 hours preoperatively and on postoperative day 2
  Patients will be evaluated by echocardiography 24 hours preoperatively and on postoperative day 2, and TAPSE will be recorded in millimeters (mm).
Echocardiographic Assessment: Pulmonary Artery Pressure (PAP) | 24 hours preoperatively and on postoperative day 2
  Patients will be evaluated by echocardiography 24 hours before surgery and on the second postoperative day, and PAP will be recorded in millimeters of mercury (mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Ankara, yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No